CLINICAL TRIAL: NCT03357133
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of Early Administration of Tirofiban in Acute Ischemic Stroke Patients Treated With Intravenous Alteplase Thrombolysis
Brief Title: Tirofiban for Patients Treated With Alteplase
Acronym: MR TEA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The number and speed of enrollment were significantly less than expected.
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017032
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban and alteplase (Experimental)
  Interventions: Drug: Tirofiban
- Alteplase (Placebo Comparator)
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tirofiban — Tirofiban Injection after the alteplase intravenous thrombolysis
  Arms: Tirofiban and alteplase
Drug: Alteplase — Only alteplase intravenous thrombolysis
  Arms: Alteplase

SUMMARY:
After intravenous thrombolysis, the overall recanalization rate is 46%, and recclusion after initial recanalization occurs in 14-34%. In the MR TEA, the investigators compared the effects of administration of tirofiban in acute ischemic stroke patients treated with intravenous alteplase thrombolysis with alteplase alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Ischemic stroke symptom with onset ≤4.5 hours treated with IV rt-PA according with local guidelines.
* 6≤ NIHSS ≤20 before IV tPA, or NIHSS >20 but decrease ≥ 8 after IV rt-PA.
* ≥ 4 point total NIHSS or ≥ 2 point in one NIHSS category during and after the IV rt-PA compared to immediately before worsening, an emergency CT scan should be performed to exclude intracranial hemorrhage
* Patients or their legally acceptable representative agreed to the treatment and signed the informed consent form

Exclusion Criteria:

* Patients whom the treating physician is planning to treat with mechanical thrombectomy or other endovascular procedure (e.g. Intra-arterial thrombolysis) according with local guidelines.
* Patients had used antiplatelet therapy in the past 5 days before the stroke.
* Patients had used anticoagulant therapy in the past 5 days before the stroke.
* Scheduled for surgery or interventional treatment requiring study drug cessation.
* CT scan finding of hypoattenuation involving ≥1/3 of the MCA territory.
* Any evidence of clinically significant bleeding ,or known coagulopathy.
* Renal insufficiency (creatinine clearance rate <30ml/min)
* Hepatic dysfunction (ALT >2 folds of Upper limit of normal value or AST>2 folds of Upper limit of normal value).
* Pre-existing disability with ≥ mRS 2.
* Known allergic to tirofiban or other glycoprotein IIb/IIIa antagonist.
* Severe non-cerebrovascular disease with life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The rate of favorable outcome | 90 days
  favorable outcome was defined as a score of 0, or 1 on the modified Rankin scale

SECONDARY OUTCOMES:
mRS ≤2 | 90 days
NIHSS score | 7 days
Deterioration after improvement | 24 hours
Final infarct size | 24 hours

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage | 7 days or discharge
Severe systemic bleeding | 7 days or discharge
Stroke-related death | 90 days
Death form any cause | 90 days

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Suzhou Municipal Hoapital, Suzhou, Anhui
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Central Hospital of Luohe City, Luohe, Henan
  - Luzhou People's Hospital, Luzhou, Sichuan
  - Xiangtan Central Hospital, Xiangtan
  - The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou